CLINICAL TRIAL: NCT03609125
Title: Cord Blood Serum in the Treatment of Neuro-Degenerative Ophthalmic Diseases. 1-Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Luigi Fontana, Full Professor of Ophthalmology - University of Bologna, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOBologna
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Glaucoma; Neuro-Degenerative Disease
Keywords: cord blood; neuroprotection; growth factors
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBS eyedrop (Experimental): The product is prepared from cord blood serum (CBS) analyzed in advance with regard to the content of specific neurotrophic growth factors.
  Interventions: Other: CBS eyedrop

INTERVENTIONS:
Other: CBS eyedrop — The product is dispensed as sterile frozen vials containing 0.8 ml of product for the daily administration. The product is thawed and administered at a dose of 1 drop / 8 times each eye during the waking period.

SUMMARY:
A non-randomized, monocentric clinical study with a four month follow-up period , using a cord blood serum (CBS) eye drops in glaucoma patients. The purpose of the study analyzes whether the addition of CBS to hypotonic therapy is able to slow down the progression of anatomical and functional damage induced by glaucoma. The study evaluates the differences after two months of treatment as compared to baseline and after two-month from the end of the treatment.

DETAILED DESCRIPTION:
The treatment of neuroprotection of degenerative ophthalmological diseases is currently proposed by administering products belonging to the category of food supplements (nutraceuticals containing amino acids and vitamins) or compounds of vegetable origin (Curcumin, flavonoids taken with food consumption of apples and oranges, LBP Polysaccharides from goji berries etc) or specific synthesis molecules (Memantine, Citicoline, Brimonidine, Omotaurina, Polyphenols).

The rationale for the use of eye drops prepared from the blood, and in particular Cord Blood Serum (CBS), as a source is mainly based on its content in growth factors (Growth factors, GF). with particular reference in neurotrophic GFs .

Enrollment of 20 patients with glaucoma and documented progressive retinal ganglion cells (RGC) dysfunction and degeneration was performed. The product to be administered was analyzed with respect to the levels of BDNF (Brain Derived Neurotrophic Factor), beta-NGF (Neural Growth Factor) , GDNF (Glial Derived Neuronal Factor), and EGF (Epidermal Growth Factor).

Functional, electro-physiological, and structural parameters were evaluated at baseline, after two months of treatment, and after two months from the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to join the study (all eligibility criteria must be met at the screening and baseline visits unless otherwise noted):

1. Participant must be medically able to undergo the testing required in the schedule of visits
2. Participant's clinical diagnosis must be consistent with glaucoma, characterized by the following features:

   1. Clinical evidence of progressive retinal ganglion cell (RGC) dysfunction and degeneration using both visual field and at least one structural modality as established by: i. Glaucomatous visual field abnormality. ii. Mean deviation (MD) of -3 to -15 dB. iii. Minimum average retinal nerve fiber layer (RNFL) thickness of 60 μm and maximum average RNFL of 90 μm.
   2. Residual visual field preservation including best-corrected visual acuity (BCVA) better than 20/200 in both eyes.
3. Participant's glaucoma must be clinically stable, with intraocular pressure (IOP) < 21.

Exclusion Criteria:

1. Participant has other optic nerve or retinal degenerative disease causing vision loss, irrespective of whether it is currently treated or untreated.
2. Participant is blind in one eye;
3. Participant has optic nerve atrophy
4. Participant is receiving systemic steroids or immunosuppressive drugs, or is on chemotherapy
5. Participant has a history of ocular herpes zoster.
6. Participant has uveitis or other ocular inflammatory disease.
7. Participant has a requirement of acyclovir
8. Participant has evidence of corneal opacification or lack of optical clarity.
9. Participant has diabetic macular edema and/or diabetic retinopathy.
10. Participant has a history of malignancy
11. Participant is pregnant or lactating.
12. History of use of drugs with known retinal toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
IOP (Intraocular pressure) | baseline, after two months of treatment, after two months from end of treatment
  Change of IOP at baseline, after treatment , and after two months from the end of treatment

SECONDARY OUTCOMES:
BCVA (Best corrected visual acuity) | baseline, after two months of treatment, after two months from end of treatment
  The change in best corrected visual acuity (BCVA) through baseline, 2 and 4 months from end of treatment
Visual Field | baseline, after two months of treatment, after two months from end of treatment
  Evaluation of change in visual field 24-2 and 10-2, through baseline, 2 and 4 months as assessed by any one of the following two indices:
  1. Pattern Standard Deviation (PSD);
  2. Mean Deviation (MD).
Fundus ophthalmoscopy | baseline, after two months of treatment, after two months from end of treatment
  Ophthalmoscopy of the following structures - Optic nerve - Choroid - Retina / Macula - Vitreous - Cup / Disco ratio performed by fundus oftlamoscopy
Structural measure of retinal nerve fiber layer thickness | baseline, after two months of treatment, after two months from end of treatment
  The change in retinal nerve fiber layer thickness as measured by spectral domain optical coherence tomography (sdOCT).
ERG (Electroretinogram) | baseline, after two months of treatment, after two months from end of treatment
  PERG: obtained with low temporal frequencies (maximum 4 hz equivalent to 8 inversions per second). Reversal rate: 2 hz (4 inversions / sec). Contrast: ceiling for white and black squares. Luminance: photopic. Wave width P50-N95 and wave latency P50.
  Flash ERG: ERG 3.0 - maximal response in the eye adapted to the dark. Full-field stimulation with Ganzfeld's dome. Amplitude A1-B1 (the amplitude of the wave b is measured from the peak of the wave until to the peak of the wave b) - the latency of the wave b is measured by the flash lighting at the peak of the wave b

CONTACTS AND LOCATIONS:
Overall Officials: Luigi FONTANA, MD, PhD, Principal Investigator — AOU Policlinico S.Orsola-Malpighi and Alma Mater Studiorum University of Bologna
Locations (1):
- IRCCS AOUBO, Ophthalmology Unit, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
data will be published in a scientific manuscript